CLINICAL TRIAL: NCT06000553
Title: Early Detection of Pancreatic Cancer in Patients With Papillary and Mucinous Intracanal Tumours of the Pancreas Papillary and Mucinous Tumours of the Pancreas PCS-IPMN-IPC 2023-005
Brief Title: Early Detection of Pancreatic Cancer in Patients With Papillary and Mucinous Intracanal Tumours of the Pancreas Papillary and Mucinous Tumours of the Pancreas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PCS-IPMN-IPC 2023-005
Record Dates: First submitted 2023-06-13; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: PAPILLARY AND MUCINOUS INTRACANAL TUMORS OF THE PANCREAS

STUDY DESIGN:
Intervention Model Description: the patient takes specific blood samples for the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collection of blood and tumor samples (Other)
  Interventions: Other: blood sampling at inclusion, 6 months, 1 year and 2 years. Tumor and intracystic fluid samples are taken only if a biopsy is planned following MRI results.

INTERVENTIONS:
Other: blood sampling at inclusion, 6 months, 1 year and 2 years. Tumor and intracystic fluid samples are taken only if a biopsy is planned following MRI results. — If the patient agrees to take part in the study, he or she will have a blood sample taken from 8 x 4 ml EDTA tubes at the time of inclusion in the trial.Then, at 6 months (+/- 1 month), 1 year and 2 years, the patient will have the same blood sample as at inclusion.If a biopsy is performed as part of routine care, a tumor sample will be taken and sent to the IPC pathology department for FFPE block. If a biopsy is performed and the patient consents, a cystic fluid sample will be taken.

SUMMARY:
This trial is a prospective, exploratory and descriptive study. The primary objective is to identify early diagnostic biomarkers in patients with TIPMP based on the analysis of Treg lymphocyte subpopulations and epigenetic signatures, and the secondary objective is to characterize the biological processes underlying the transformation of a pre-neoplastic lesion into established ADPC.

DETAILED DESCRIPTION:
To meet the objectives of the study, patients will have blood samples taken at the time of their TIPMP monitoring, i.e. at inclusion, 6 months, 1 year and 2 years. If echo-endoscopy is performed during MRI monitoring of their disease, and a sample is taken as part of the treatment, a tumor sample and an intra-cystic fluid sample will be collected as part of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18
2. Patient with intermediate-risk or high-risk TIPMP according to the European Study Group on Cystic Tumours of the Pancreas (3)
3. Signed consent to participate
4. Affiliation with a social security scheme, or beneficiary of such a scheme.

Exclusion Criteria:

1. Pregnant or breast-feeding woman
2. Person in an emergency situation or unable to give consent.
3. Adult subject to a legal protection measure (adult under guardianship, curatorship or safeguard of justice),
4. Unable to undergo medical follow-up for geographical, social or psychological reasons.
5. contraindication to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
the aim is to search for immune and metabolic abnormalities in patients with at-risk TIPMP in the blood or by echo-endoscopic sampling, then compare and combine them with the criteria used in clinical practice. | for two years
  Biomarkers will be studied to determine whether those selected have been effective in identifying patients with pancreatic adenocarcinoma.

IPD SHARING:
Plan to Share IPD: Undecided